CLINICAL TRIAL: NCT05650463
Title: Evaluation of a Smartphone-based Screening Tool (Picterus Jaundice Pro) for Neonatal Jaundice in Dark Skin Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Stockholm
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): There is only one arm in this study which is to enable high qualitative estimation of bilirubin levels in the blood of new-borns with darker skin types using Picterus JP.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place.

SUMMARY:
A cross-sectional study at the Södersjukehuset facility (Stockholm, Sweden) collect data of newborns from a population with Neomar scale type 4 to adjust the algorithm of Picterus JP

DETAILED DESCRIPTION:
To adjust Picterus JP to work in newborns with more pigmented skin, the investigators will collect a data set at Sachsska barnsjukhuset Södersjukhuset, Stockholm Sweden from 150 newborns with dark skins using Picterus JP, TcB, skin measurements from a spectrometer, visual assessment, and total serum bilirubin (TSB) levels. As a control, newborns with Neomar scale 1-3 will be included.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age ≥ 37
* Birth weight ≥ 2500g
* Age 1 - 14 days
* Will have a blood sample performed, either for clinically suspected jaundice or newborn screening sample

Exclusion Criteria:

* Infants showing signs of inborn disease
* Infants transferred to pediatric ward for treatment
* Infants that have received phototherapy

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in newborns, independent of skin color, using Picterus JP | 6 months
  Evaluate of smartphone-based screening tool (Picterus JP) for neonatal jaundice in newborns with Neomar neonatal skin color scale type 4 (with type 1 being lower-melanin level and Type 4 being higher-melanin level)

SECONDARY OUTCOMES:
Comparison of Picterus-generated estimate with TsB | 1-2 hours
  Compare bilirubin estimates calculated with the adjusted algoritm from the images with TSB measurements
Comparison of Picterus-generated estimate with TcB | 5-10min
  Compare bilirubin estimates calculated with the adjusted algoritm from the images with TcB measurements
Comparison of Picterus-generated estimate with visual assessment. | 5-10min
  Compare bilirubin estimates calculated with the adjusted algoritm from the images with visual assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lobke Gierman, PhD, Principal Investigator — Picterus AS
Locations (1):
- Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No